CLINICAL TRIAL: NCT01480206
Title: 3D Interventional Tools for Endovascular Procedures in the OR
Brief Title: Overlay of 3D Scans on Live Fluoroscopy for Endovascular Procedures in the Hybrid OR
Status: Completed | Type: Observational
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Other Study IDs: XCY611-110165
Record Dates: First submitted 2011-11-23; First posted 2011-11-28 (Estimated); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Abdominal Aortic Aneurysm (AAA); Thoracic Aortic Aneurysm (TAA); Carotid Stenosis; Visceral Artery Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aortic Aneurysm, Thoracic; Carotid Stenosis | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Endovascular Aortic Repair (EVAR) — Use of 3D interventional imaging tools in endovascular procedures in the surgical environment
  Other Names: EVAR, TEVAR

SUMMARY:
As endovascular procedures become more complex, there is a growing need for 3D image overlay to assist with device guidance and placement. Currently, a 3D image is typically created intra-operatively using 3D rotational angiography (3D-RA) or cone-beam CT (XperCT). This 3D image may then be overlaid on live fluoroscopy to provide 3D guidance information (Dynamic 3D Roadmapping). Philips Healthcare multimodality overlay products allows registration of a pre-acquired MR/CT or 3D rotational image to live fluoroscopy.

DETAILED DESCRIPTION:
Endovascular treatment is performed under the guidance of an X-ray angiography system. Fluoroscopy and conventional 2D digital subtraction angiography (DSA) are used to navigate the interventional device (and implant) across the lesion to achieve a correct bridging of the diseased region of the vessel, while excluding the involvement of patent vessels. Drawbacks of these peripheral interventions include the radiation dose, use of contrast, and need for a clinician with excellent wire-handling skills. The use of 2D imaging alone may not be enough to describe the three-dimensional(3D) relationship between interventional devices (and implants) and the complex vascular anatomy, often making positioning, deployment and evaluation suboptimal. In addition, the endovascular approach can lead to complications such as in-stent thrombosis and type II endoleak (in the case of aortic aneurysms) for which 2D imaging along is again sub-optimal for re-intervention planning and guidance.

As endovascular procedures become more complex, there is a growing need for 3D image overlay to assist with device guidance and placement. Currently, a 3D image is typically created intra-operatively using 3D rotational angiography (3D-RA) or cone-beam CT (XperCT). This 3D image may then be overlaid on live fluoroscopy to provide 3D guidance information (Dynamic 3D Roadmapping). 3D navigation can also be acquired by registration of a pre-acquired MR/CT or 3D rotational image to live fluoroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age 18-90, of both genders and all races
* Patients undergoing elective AAA or TAA repair or carotid stenting or peripheral intervention
* Patients already selected for endovascular treatment by preoperative CT angiogram
* Patients with preoperative CT performed within 4 months of operation

Exclusion Criteria:

* Patients refusing or incapable of providing informed consent
* Patients undergoing emergent or ruptured AAA repair
* Patients with known connective tissue disorders
* Patients with aortic dissections
* Patients participating in other EVAR, IDE, or IND trials
* Patients with anticipated adjunctive intervention requiring additional intravenous contrast
* Patients with anticipated endograft extension distal to the common iliac artery
* Patients without CT angiogram performed at BIDMC with standard EVAR protocol
* Patients without CT angiogram performed within 4 months of operation
* Patients with glomerular filtration rate (GFR) < 60 mL/min/1.73m2
* Patients with contraindication to intravenous contrast
* Patients with disability or previous implants precluding adequate visualization on rotational imaging

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with age 18-90, of both genders and all races Patients undergoing elective AAA or TAA repair or carotid stenting or peripheral intervention Patients already selected for endovascular treatment by preoperative CT angiogram Patients with preoperative CT performed within 4 months of operation
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2011-09-13 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
feedback to improve the usability of the Vessel Navigator | one month after procedure
  PI answers questions to help improve the usability of the VesselNavigator

CONTACTS AND LOCATIONS:
Overall Officials: Marc Schermerhorn, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States